CLINICAL TRIAL: NCT02312583
Title: Efficacy the Online Program iFightDepression for the Treatment of Mild and Moderate Depression
Brief Title: Efficacy of an Online Program for the Treatment of Mild and Moderate Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Víctor Pérez, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: iFightDepression
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Depression
Keywords: depression; cognitive-behavior intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychoeducational online information (Sham Comparator): Psychoeducational online information. During 7 weeks as a complement to the usual treatment.
  Interventions: Behavioral: Psychoeducational online information
- iFightDepression online programme. (Experimental): iFightDepression online programme. During 7 weeks as a complement to the usual treatment.
  Interventions: Behavioral: iFightDepression online programme

INTERVENTIONS:
Behavioral: Psychoeducational online information — Psychoeducational online information. During 7 weeks as a complement to the usual treatment. Participants will have access to online psychoeducational material for depression.
  Arms: Psychoeducational online information
Behavioral: iFightDepression online programme — iFightDepression online programme. During 7 weeks as a complement to the usual treatment.
  Participants will complete the modules of a structured online programme for depression
  Arms: iFightDepression online programme.

SUMMARY:
iFighDepression is an online self-help programme based on cognitive-behavioral therapy that could be useful for the treatment of mild to moderate depression

DETAILED DESCRIPTION:
Major depression (MD) is a disease with a great impact on people´s functioning and is the second leading cause of disability worldwide. It is a condition with a high prevalence, about 10% of men and 20% of women in the population will be diagnosed MD throughout their lives, and has an effect on high economic costs to health services.

While there are many effective therapeutic options for the treatment of depression, many people with depressive episodes do not receive an appropriate treatment or, in fact, do not receive any treatment at all. The social stigma, difficulties to access mental health services, to integrate therapy sessions into working life, or problems to pay for treatment are some of the main barriers to receive adequate treatment.

On-line interventions are easily accessible and low cost, and different studies suggest that these interventions have significant and lasting improvements in different mental disorders. These studies indicate that this type of treatment would be indicated for disorders that, as the case of MD, have a high prevalence and relatively low help-seeking for treatment.

iFighDepression is an online self-help programme for mild to moderate depression that has been developed in the context of the European project Preventing Depression and Improving Awareness through Networking in the European Union (PREDI-NU) which is managed by the European Alliance Against Depression (EAAD). It involves the most complete integration of the cognitive-behavioral online programs available to date, which is a format of intervention that has been proven effective in reducing depressive symptoms in several randomized controlled trials. IFightDepression is currently in pilot phase in 7 European Union countries, including Spain.

The purpose of this project is to study the therapeutic effect of the iFightDepression online programme in patients with mild to moderate depression

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder according to Diagnostic and Statistical Manual (DSM-IV-TR) criteria.
* Clinical severity between mild and moderate (according to ICG severity scale).
* A minimum of reading comprehension and knowledge of internet browsing.
* Availability to access internet during the 7 weeks of the intervention.
* Informed written consent provided.

Exclusion Criteria:

* Suicidal ideation (assessed by the HDRS and clinical interview).
* Presence of delusional ideas or hallucinations, consistent or not with the mood.
* Other concomitant psychiatric pathologies of the Axis I or Axis II according to Diagnostic and Statistical Manual (DSM-IV-TR) at the time of entry to the study.
* To be currently enrolled in a structured programme/treatment of psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in depression Scale | From baseline to 7 weeks
  Efficacy will be assessed by using the Hamilton Depression Scale, version 17 items (HDRS-17). The HDRS-17 will be administered at baseline, 4 weeks and 7 weeks.

SECONDARY OUTCOMES:
Change in the Clinical Global Impression of Severity and Improvement | From baseline to 7 weeks
  Clinical Severity will be assessed using the Scale of Clinical Global Impression of Severity and Improvement (ICG-s and ICG-m). Hetero and Self-Administered versions.
  Scale of Clinical Global Impression of Severity and Improvement (ICG-s) at baseline. and at 7 weeks Scale of Clinical Global Impression of Severity and Improvement (ICG-m) at baseline and at 7 weeks.
Change in depressive symptomatology | From baseline to 7 weeks
  Depressive symptomatology measured by the Self-Report Patient Health Questionnaire-9 (PHQ-9). Measure will be done once a week.
Change in the Remission from Depression | From baseline to 7 weeks
  Remission from Depression Questionnaire (RDQ): Self-Report in relation to different domains considered as relevant by the patients themselves in defining the construct of remission in the scope of depressive disorders. Measure will be done once a week.
Change in quality of life | From baseline to 7 weeks
  Change measured using the EuroQoL Quality of Life Scale (EQ-5 d). It is a Self-Report measure of health variables which is commonly used as an indicator of quality of life.
Change in functional impairment | From baseline to 7 weeks
  Functional impairment assessed by using the Functioning Assessment Short Test (FAST). It evaluates the functional impairment in patients suffering from mental illness, including the Major Depression.
Users satisfaction score | One measure at 7 weeks
  User´s satisfaction by using the Satisfaction Questionnaire: a questionnaire of satisfaction used in the validation of the programme iFightDepression within the project PREDI-NU. It includes questions about the manageability of the programme and the beneficial aspects perceived by the user.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Perez, MD, PhD, Principal Investigator — Institute of Neuropsychiatry and Addictions (INAD). Parc de Salut Mar, Hospital del Mar
Locations (5):
- Spain (5):
  - Institute of Neuropsychiatry and Addictions (INAD). Parc de Salut Mar, Hospital del Mar. Passeig Maritin, 25-29., Barcelona, Barcelona
  - Hospital de Sant Pau de Barcelona. Department of Psychiatry. Servicio de Psiquiatria. Carrer de Sant Quintí, 89, Barcelona
  - Red de Salud Mental de Guipúzkoa (Guipuzcoan Mental Health Network). Pº Dr.Begiristain, 115 (Aránzazu building)., Donostia / San Sebastian
  - Hospital Universitario de la Princesa. Department of Psychiatry. Calle de Diego León, 62, Madrid
  - Hospital Parc Taulí de Sabadell. Community Mental Health Services. Parc Taulí 1,, Sabadell

REFERENCES:
- [Derived] Justicia A, Elices M, Cebria AI, Palao DJ, Gorosabel J, Puigdemont D, de Diego-Adelino J, Gabilondo A, Iruin A, Hegerl U, Perez V. Rationale and methods of the iFightDepression study: A double-blind, randomized controlled trial evaluating the efficacy of an internet-based self-management tool for moderate to mild depression. BMC Psychiatry. 2017 Apr 19;17(1):143. doi: 10.1186/s12888-017-1306-2. PMID 28420367